CLINICAL TRIAL: NCT03573791
Title: Identification of Tissue Biomarkers for Predicting Neoadjuvant Chemoradio-resistance in Patients With Middle-low Local Advanced Rectal Cancer.
Brief Title: Biomarkers for Predicting Neoadjuvant Chemoradio-resistance for Middle-low Advanced Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zheng Wang, MD/PhD, Study chair, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: WHUHGE-R01
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer; Cancer of Rectum; Cancer of the Rectum; Neoplasms, Rectal; Rectal Tumors; Rectum Cancer; Rectum Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor biopsy samples are collected before neoadjuvant therapy when participants undergo colonoscopy or endoscopic ultrasonography. Two pieces of tumor tissue specimens will be extracted. These tissues will be stored at the tumor specimen bank and gene expression profile of these tumor samples will be analyzed using RNA sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete response: After neoadjuvant therapy, postoperative pathological examination will be performed to evaluate the efficacy of the therapy. Define postoperative staging ypT0N0 as complete response.
- Poor response: After neoadjuvant therapy, postoperative pathological examination will be performed to evaluate the efficacy of the therapy. Define postoperative staging >ypT1-2N0 as poor response.

SUMMARY:
Neoadjuvant therapy has been widely applied to locally advanced rectal cancer. However, about 50% of patients receiving this therapy do not respond well as evidenced by the fact that their T or N stages are not effectively decreased judged by postoperative pathological examination. The purpose of this trail is to identify the biomarkers (from within patients' tumor mass before neoadjuvant therapy) to predict resistance to neoadjuvant therapy. These biomarkers can help stratify neoadjuvant-resistant patients towards surgery while avoiding unnecessary chemoradio-based neoadjuvant therapy.

DETAILED DESCRIPTION:
According to postoperative pathological examination results, all participants will be divided into two groups: complete response (ypT0N0) and poor response (>ypT1-2N0). Differentially expressed genes between complete response and poor response will be analyzed. A scoring formula will be established based on the results. Tumor tissue samples are collected before neoadjuvant therapy and will be analyzed via RNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology proved to be adenocarcinoma of the rectum.
* The edge of tumor is within 12cm of anus margin.
* According to the eighth edition of AJCC TNM staging standard ,that staging for Ⅱ-Ⅲ period, as T3-T4, N0 or any T, N1-2.
* There is no history of chemotherapy, radiotherapy or immunotherapy before neoadjuvant therapy.
* Understand and agree to sign the informed consent for the study.

Exclusion Criteria:

* With intestinal obstruction or impending obstruction, or perforation.
* With other malignancies occurred within 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from Wuhan Union Hospital or Hubei Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Comparing gene expression differences between poor response group and complete response group by using RNA sequencing. | 6 months
  Using RNA-seq sequencing method to obtain the whole genome transcription profiles of the poor response group and complete response group, and compare the gene expression differences between these two groups.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The total survival time of the participants from joining the group to the death. If the death time is unknown, the relevant participants will be excluded for analysis.
Progression Free Survival(PFS) | 3 years
  The time period that from participants joining the groups to the progression of disease(recurrence or metastasis) or death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, MD/PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang GJ, Park IJ, You YN, et al. Neoadjuvant treatment response and outcomes in locally advanced rectal cancer: Establishing oncologic benchmarks. Journal of Clinical Oncology 29(15):3545-3545,2011.